CLINICAL TRIAL: NCT05851326
Title: A Combination of Low-Energy Ultrasound, Electrical and Magnetic Field Stimulation in Patients With Therapy-Resistant Myofascial Pain Syndrome: A Randomized, Controlled, Double-Blind Multi-Center Study
Brief Title: Low-Energy Ultrasound, Electrical and Magnetic Field Stimulation in Therapy-Resistant Myofascial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sobet AG (Industry)
Collaborators: Klinikum Klagenfurt am Wörthersee (Other); Krankenhaus der Elisabethinen Graz (Unknown); Krankenhaus St. Vinzenz Zams (Unknown); La Tour Hospital (Other); Schmerzklinik Zürich (Unknown); Salem-Spital Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sonodyn
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Myofascial Pain Syndrome - Lower Back; Myofascial Pain Syndrome - Neck; Myofascial Pain Syndrome - Tension Headache
Keywords: Myofascial Pain Syndrome; Low-Energy Stimulation; Ultrasound, Electrical and Magnetic Field Stimulation; Transcutaneous Pain Therapy; Chronic Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Sonodyn Therapy (Treatment Group) (Experimental): Patients will remain on treatment for 3 weeks and will activate their device 3 times a day for 10 minutes each.
  Interventions: Device: Active Sonodyn
- Sham Therapy (Control Group) (Sham Comparator): Patients will remain on sham treatment for 3 weeks and will activate their device 3 times a day for 10 minutes each.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Active Sonodyn — Sonodyn emits ultrasound, electrical and magnetic stimulation signals with a pre-defined, fixed set of parameters for each of the independently operated power sources.
  Arms: Active Sonodyn Therapy (Treatment Group)
Device: Sham — Non-functional Sonodyn device that cannot convey any energy signals to the device output, however, looks and behaves fully identical as the active Sonodyn device.
  Arms: Sham Therapy (Control Group)

SUMMARY:
Sonodyn is an investigational device that within this clinical investigation is intended for use in patients suffering from low back pain, tension headache or neck pain, originating from therapy-resistant myofascial pain syndrome.

Myofascial pain syndrome is a prevalent pain condition in the adult population and a common cause of pain and dysfunction in the musculoskeletal system. It is a trigger point-induced regional musculoskeletal pain disorder affecting one or more muscles or groups of muscles.

Sonodyn is a handheld medical device that combines low-energy ultrasound, electrical and magnetic field stimulation for non-invasive transcutaneous treatment of chronic myofascial pain syndrome. Sonodyn is a battery-operated, rechargeable stimulation device to be placed over specific trigger points for associated pain patterns in the human body. It emits ultrasound, electrical and magnetic stimulation signals with a pre-defined set of parameters for each of the independently operated power sources.

The study will follow a prospective, randomized, sham-controlled, double-blind parallel group design. It will be conducted as a multi-center investigation at 6 sites in Austria and Switzerland. Patients are randomized in a 2:1 ratio into Treatment and Control.

* Active Sonodyn therapy (Treatment)
* No therapy (Sham Control)

Two types of Sonodyn devices will be used: a fully functional one for Therapy arm patients that can deliver stimulation, and a non-functional one for Control arm patients that cannot convey any energy signals to the device output. The devices will look fully identical.

Randomization will be stratified by study site, pain diagnosis and sex of the patient.

For each subject, after a screening phase of 1 week, patients will be treated for 3 weeks with a follow-up of additional 8 weeks, adding up to 12 weeks. During treatment patients will activate their device 3 times a day for 10 minutes each.

During screening, treatment and follow-up period, all patients will twice per day report the average and maximum intensity of their pain Numeric Rating Scale (NRS). Patients will also enter the date, amount, and time of intake of rescue medication, if applicable.

The primary objective of this study is to assess the impact on pain. Secondary objectives are to compare the performance between active therapy and sham, as well as to correlate changes in pain intensity with other pain related scales.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 99 years at screening
* Patient has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures
* Patient is suffering from one of the following chronic pain conditions originating from myofascial pain:

  * low back pain
  * tension headache
  * neck pain

having been persisting for a minimum of 3 months and where myofascial pain syndrome is the pre-dominant cause for pain.

* Patient is constant with respect to pain treatment for 1 week during the screening phase
* A daily average NRS >= 4 on 4 out of 7 days in the screening phase
* Compliance with the daily status reporting requirements as demonstrated

Exclusion Criteria:

* Patients with active implants
* Allergy against rescue medication used during the study
* Pregnancy
* Mental or physical impairments that represent a source of risk for handling the device
* Patients with cerebral spams (epilepsy)
* Patients with psychiatric diseases or somatoform pain disorders
* Patients with oral morphine equivalent of more than 120mg daily dose
* Patients taking centrally acting muscle relaxants like Sirdalud or benzodiacepines
* Patients with a contraindication against NSAID's
* Presence of artificial joints made from methylmethacrylate or polyethylene at stimulation site
* Presence of ferromagnetic metal implants at stimulation site, especially aneurysm clips, dental implants, etc.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Average Numeric Rating Scale (NRS) | 3 weeks
  Change in Treatment group from Baseline to EoT in average Numeric Rating Scale (NRS, 0-10, with 0 indicating no pain and 10 indicating the worst pain that the patient had ever experienced) per day

SECONDARY OUTCOMES:
Difference in average NRS between groups - Baseline to EoT | 3 weeks
  Difference between groups in change of average NRS from Baseline to EoT
Maximum NRS - Baseline to EoT | 3 weeks
  Change from Baseline to EoT in maximum NRS in both groups
Average and maximum NRS - Baseline to end of follow-up | 11 weeks
  Change from Baseline to end of follow-up in average and maximum NRS in both groups
AUC of average and maximum NRS - Baseline to EoT | 3 weeks
  Baseline-adjusted area under the curve (AUC) of average and maximum NRS from Baseline to EoT in both groups
Average and maximum NRS - Follow-up | 8 weeks
  Average and maximum NRS during follow-up in both groups
Medication consumption | 11 weeks
  Pain and rescue medication consumption during treatment and follow-up phase in both groups
EQ-5D-5L | 11 weeks
  EQ-5D-5L questionnaire from Baseline to EoT and end of follow-up
Quality of sleep | 11 weeks
  Quality of sleep questionnaire from Baseline to EoT and end of follow-up
Socioeconomic data | 4 weeks
  Change in socioeconomic data from Screening to EoT

OTHER OUTCOMES:
Safety Outcome #1 | 3 weeks
  Adverse Events (AEs), Adverse Device Effects (ADEs), and Device Deficiencies (DDs) observed until EoT
Safety Outcome #2 | 11 weeks
  Serious Adverse Events (SAEs), Serious Adverse Device Effects (SADEs), and related AEs observed until end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Likar, Prof. Dr., Principal Investigator — Klinikum Klagenfurt am Wörthersee
Locations (6):
- Austria (3):
  - Schmerzambulanz, Krankenhaus der Elisabethinen Graz, Graz
  - Abteilung für Anästhesiologie und Intensivmedizin, Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Krankenhaus St. Vinzenz Zams, Zams
- Switzerland (3):
  - RSB Neurochirurgie AG, Salem-Spital Bern, Bern
  - Clinique de la Douleur, La Tour Hospital, Meyrin
  - Schmerzklinik Zürich AG, Zurich

IPD SHARING:
Plan to Share IPD: No